CLINICAL TRIAL: NCT00357149
Title: Randomized Phase II Trial of Neoadjuvant Docetaxel Plus Cisplatin and 5-fluorouracil Followed by Concomitant Chemoradiotherapy and Chemoradiotherapy Alone in Patients With Locally Advanced Squamous Cell Carcinoma of the Head and Neck.
Brief Title: Neoadjuvant Docetaxel Plus Cisplatin and 5-fluorouracil (TPF) Followed by Concomitant Chemoradiotherapy and Chemoradiotherapy Alone in Locally Advanced Squamous Cell Carcinoma of the Head and Neck Patients (SCCHNS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XRP6976F_2501
Record Dates: First submitted 2006-07-26; First posted 2006-07-27 (Estimated); Last update posted 2009-12-07 (Estimated); Status verified 2009-12

CONDITIONS: Head and Neck Neoplasms
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Docetaxel; Cisplatin; Fluorouracil; Radiotherapy

ARMS (2):
- A (Active Comparator): Cisplatin from day 1 to day 4 and 5-FU for 4 days starting immediately after the end of cisplatin infusion on day 1. Both drugs were administered during week 1 and 6 of irradiation, starting from day 1 of weekly radiotherapy.
  Interventions: Drug: Concomitant cisplatin, 5-FU and radiotherapy
- B (Experimental): Docetaxel followed by cisplatin and 5-FU from day 1 to day 4 starting after the end of cisplatin infusion. The cycle was repeated every 3 weeks up to a total of 3 cycles. After 3-6 weeks from the end of neoadjuvant chemotherapy, patients will receive with the same modality of arm A (reference arm).
  Interventions: Drug: Docetaxel, cisplatin and 5-FU treatment followed by concomitant cisplatin, 5-FU and radiotherapy

INTERVENTIONS:
Drug: Docetaxel, cisplatin and 5-FU treatment followed by concomitant cisplatin, 5-FU and radiotherapy
  Arms: B
Drug: Concomitant cisplatin, 5-FU and radiotherapy
  Arms: A

SUMMARY:
To evaluate the rate of clinical complete response 6-8 weeks after treatment with docetaxel plus cisplatin and 5-fluorouracil followed by chemoradiotherapy and after chemoradiotherapy alone in patients with locally advanced squamous cell carcinoma of the head and neck.

ELIGIBILITY:
Inclusion criteria:

* Histologically or cytologically proven squamous cell carcinoma of the head and neck.
* Primary tumor sites eligible: oral cavity, oropharynx, hypopharynx. Although they are admittedly of squamous cell types, the following tumors will be excluded because of theY responsiveness to chemotherapy: tumors of the nasal and paranasal cavities, larynx and of the nasopharynx.
* Stage III or IV disease without evidence of distant metastases verified by chest X Ray and/or lung CT scan, abdominal ultrasound, or CT (liver function test abnormalities); bone scan in case of local symptoms.
* At least one measurable lesion.
* Tumor considered inoperable after evaluation by a multidisciplinary team (i.e. a surgeon, a medical oncologist and a radiation oncologist).
* No previous chemotherapy or radiotherapy for any reason and no previous surgery for squamous cell carcinoma of the head and neck patients (other than biopsy) are allowed at time of study entry.
* Karnofsky performance status ≥ 70.
* No active alcohol addiction.
* Adequate bone marrow, hepatic and renal functions
* Patients must be available for treatment and follow-up.

Exclusion criteria

* Pregnant or lactating women or women of childbearing potential not using adequate contraception.
* Previous or current malignancies at other sites, with the exception of adequately treated in situ carcinoma of the cervix uteri, basal or squamous cell carcinoma of the skin, or other cancer curatively treated by surgery and with no evidence of disease for at least 5 years.
* Symptomatic peripheral neuropathy ≥ grade 2
* Symptomatic altered hearing ≥ grade 2
* Other serious illnesses or medical conditions including:a) Unstable cardiac disease despite treatment, myocardial infarction within 6 months prior to study entry.b) History of significant neurologic or psychiatric disorders including dementia or seizures.c) Active uncontrolled infection.d) Active peptic ulcer.e) Hypercalcemia.f) Chronic obstructive pulmonary disease requiring hospitalization during the year preceding study entry
* History of hypersensitivity reaction to polysorbate 80
* Patients requiring intravenous alimentation.
* Patients who experienced a weight loss of more than 20% of their body weight in the 3 months preceding study entry.
* Concomitant treatment with any other anticancer therapy.
* Participation in a therapeutic clinical trial within 30 days of study entry

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2003-01; Primary Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Rate of radiologic Complete Response (CR) evaluated 6-8 weeks after the completion of treatment | from end of treatment until 6-8 weeks

SECONDARY OUTCOMES:
Duration of response | from the date of first documented tumor response to the date of first documented tumor progression
Time to disease progression | From the date of the treatment start to the date of first documented progression of disease
Time to treatment failure | from the date of treatment start to the date of diagnosis of progression, withdrawal from study treatment for any reason, administration of other antitumor treatment, or death for any cause
Median length of overall survival | time interval from the date of treatment to the date of death

CONTACTS AND LOCATIONS:
Overall Officials: Georges Paizis, MD, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Milan, Italy